CLINICAL TRIAL: NCT00474773
Title: Evaluation of Post Hospital Administration of Celecoxib Following Minimally Invasive Knee Replacement Surgery: A Randomized Controlled Study
Brief Title: Evaluation of Post Hospital Administration of Celecoxib Following Minimally Invasive Knee Replacement Surgery
Status: Completed | Type: Observational
Sponsor: St. Louis Joint Replacement Institute (Other)
Collaborators: Pfizer (Industry); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: GA3190YM
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2010-01

CONDITIONS: Pain Management; Function; Minimally Invasive Total Knee Arthroplasty; Celecoxib
MeSH Terms: conditions — Agnosia | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
This study will evaluate the benefits of continuing celecoxib through six weeks of total knee arthroplasty recovery. This is a randomized, double blind study with a group of approximately 130 primary total knee patients. All patients will receive celecoxib throughout their hospitalization as per current minimally invasive total knee arthroplasty protocol. At the time of hospital discharge, participating patients will be randomly placed on either celecoxib 200mg twice a day or a placebo twice a day.

This study will determine if the continued use of celecoxib for six weeks after total knee arthroplasty hospitalization will further decrease narcotic consumption, improve knee range of motion, improve ambulatory ability, and improve patient satisfaction over patients receiving celecoxib only during the acute hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* having undergone a minimally invasive total knee by select surgeon
* voluntarily enrolled
* independent community ambulators
* only patients being discharged directly home

Exclusion Criteria:

* celecoxib allergy or intolerence
* Renal insufficiency (defined as serum creatine level >1.5 mg/dL or BUN level >22mg/dL
* History of bleeding gastic or duodenal ulceration
* New York Heart Association Class III or IV Congestive Heart Failure
* Previous myocardial infarction or cerebralvascular event
* Severe inflammatory bowel disease
* Known coagulation abnormality or hepatic disease
* Chronic coumadin administration
* Refusal by primary or cardiac physician

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: total knee canidates
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Schroer, MD, Principal Investigator — St. Louis Joint Replacement Institute
Locations (1):
- DePaul Health Center, St Louis, Missouri, United States